CLINICAL TRIAL: NCT03714152
Title: A Phase 1 Study of the Safety, Tolerability, Pharmacokinetics, and Food Effect of Single and Multiple Doses of ABI-H2158 in Healthy Volunteers; and the Multiple-Ascending Dose Pharmacokinetics and Pharmacodynamics in Patients With Chronic Hepatitis B Infection
Brief Title: A Study of ABI-H2158 in Healthy Volunteers and Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABI-H2158-101
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis B
Keywords: CHB; HBV; hepatitis B; HBeAg positive
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ABI-H2158 (Experimental): ABI-H2158 in varying doses of tablets by mouth without and with food for 1 day or 10 days
  Interventions: Drug: ABI-H2158
- Matching Placebo for ABI-H2158 (Placebo Comparator): Matching Placebo in varying doses of tablets by mouth without and with food for 1 day or 10 days
  Interventions: Drug: Placebo for ABI-H2158

INTERVENTIONS:
Drug: ABI-H2158 — 5 mg or 25 mg tablets
  Arms: ABI-H2158
Drug: Placebo for ABI-H2158 — Sugar pill manufactured to mimic the ABI-H2158 5 mg or 25 mg tablets
  Arms: Matching Placebo for ABI-H2158

SUMMARY:
This three-part, Phase 1 protocol will be the first clinical study of ABI-H2158. Parts 1 and 2 will be a Phase 1a, dose-ranging assessment of ABI-H2158 in healthy adult volunteers. If the dose-related safety, tolerability, and pharmacokinetics (PK) of ABI-H2158 in healthy volunteers are deemed satisfactory, then the study will advance to Part 3, a Phase 1b, dose-ranging assessment of ABI-H2158 in non-cirrhotic, CHB patients.

ELIGIBILITY:
Healthy volunteers:

1. Male or female between 18 and 55 years old with a BMI of 18-34 kg/m2 with a minimum body weight of 45 kg
2. Must be in good health and not have any health condition which could interfere with the absorption, distribution or elimination of study drug, or with the clinical and laboratory assessments in this study

Chronic HBV patients:

Key Inclusion Criteria:

1. Male or female ≥ 18 and ≤ 65 years of age.
2. In good general health except for chronic HBV infection, documented by:

   1. Clinical history, physical exam and routine laboratory measurements without major or clinically significant findings
   2. Serologic profile consistent with chronic HBV infection • HBeAg-positive at Screening with HBV viral load ≥ 2× 105 IU/mL
3. Liver evaluation demonstrating the absence of bridging fibrosis or cirrhosis

Key Exclusion Criteria:

1. History or evidence of decompensated liver disease at any time prior to Screening
2. History or presence of any other clinically significant current medical conditions requiring ongoing pharmacological treatment.
3. Previous treatment with any investigational HBV antiviral treatments within the last 6 months, or previous treatment at any time with an investigational HBV antiviral treatment of the same class (core protein targeted therapies).
4. Previous treatment with a commercially approved HBV therapy within the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Number of healthy volunteers and patients with chronic HBV infection with treatment-related adverse events as assessed by CTCAE v4.0. | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (14):
- United States (4):
  - Southern California Research Center, Coronado, California
  - Research and Education, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Infectious Disease Care, Hillsborough, New Jersey
- Australia (3):
  - Monash University, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- First Hospital of Jilin University, Jilin, Changchun, China
- University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong
- Auckland Clinical Studies, Auckland, New Zealand
- South Korea (3):
  - Hallym University, Chuncheon
  - Asan Medical Center, Seoul
  - Severance Hospital, Yonsei University, Seoul
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided